CLINICAL TRIAL: NCT02119507
Title: Effect of Curodont Repair in Patients With Early Approximal Carious Lesions: A Mono-centre, Controlled, Single-blinded, Randomised, Post-marketing Study
Brief Title: Effect of Curodont Repair in Patients With Early Approximal Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credentis AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P11-4-APCL
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Dental Caries
Keywords: Dental caries; Curodont Repair; P11-4
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curodont Repair (Experimental): Single application on Day 0.
  Interventions: Device: Curodont Repair
- No treatment - control (Other): No treatment as control - "wait and see".
  Interventions: Other: No treatment - control

INTERVENTIONS:
Device: Curodont Repair — Single application on Day 0
  Other Names: P11-4
  Arms: Curodont Repair
Other: No treatment - control
  Arms: No treatment - control

SUMMARY:
The purpose of this study is to evaluate the therapeutic benefit of Curodont Repair for the treatment of early approximal carious lesions compared to no treatment.

DETAILED DESCRIPTION:
All study participants must have two early approximal carious lesions in need of a treatment but not of an invasive treatment (split-mouth design). One lesion will be treated with Curodont Repair and the other will not undergo a treatment as control. Study duration is 12 months. For assessment x-ray pictures are used.

ELIGIBILITY:
Inclusion Criteria:

* Two approximal carious lesions on different teeth with at least one tooth in between
* Both study lesions must not require an invasive treatment
* Size and form of the lesions: the lesions must be fully visible and assessable on radiographs
* The two carious lesions must fall into classes:

D1 (outer half of enamel) D2 (inner half of enamel) D3 (outer part of dentine) but only if very little dentine is involved (enamel-dentine junction)

* Able and willing to observe good oral hygiene throughout the study
* Age ≥ 18 years and ≤ 65 years
* Willing and able to attend the on-study visits
* Willing and able to understand all study-related procedures
* Written informed consent before participation in the study

Exclusion Criteria:

* The two study test lesions are located on adjacent teeth
* Fluoride varnish application < 3 months prior to study treatment
* Tooth with numerous carious lesions
* Evidence of tooth erosion
* History of head and neck illnesses (e.g. head/neck cancer)
* Any pathology or concomitant medication affecting salivary flow or dry mouth
* Any metabolic disorders affecting bone turnover
* Patient suffers from diabetes
* Concurrent participation in another clinical trial
* Women who are breast-feeding, pregnant or who plan a pregnancy during the study
* Women of childbearing potential who declare being unwilling or unable to practice contraception such as hormonal contraceptives, sexual abstinence or intercourse with a vasectomised partner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Opaqueness on X-Ray | Day 360
  The primary efficacy outcome is the difference of the change in the opaqueness of the carious lesion on the x-ray picture from Day 0 to Day 365 between test and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Heimlinger, Dr. med. dent., Principal Investigator — zumstein dental clinic ag
Locations (1):
- Zumstein Dental Clinic Ag, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Brunton PA, Davies RP, Burke JL, Smith A, Aggeli A, Brookes SJ, Kirkham J. Treatment of early caries lesions using biomimetic self-assembling peptides--a clinical safety trial. Br Dent J. 2013 Aug;215(4):E6. doi: 10.1038/sj.bdj.2013.741. PMID 23969679